CLINICAL TRIAL: NCT07346703
Title: Effects of Therapeutic Exercise and Long-term Docosahexaenoic Acid (DHA) Supplementation on Physical, Physiological, Motor, Mental, and Cognitive Variables in Patients With Multiple Sclerosis.
Brief Title: Effects of DHA in Patients With Multiple Sclerosis
Acronym: DHAME
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Javier Martínez Noguera (Other)
Responsible Party: Sponsor-Investigator, Francisco Javier Martínez Noguera, Associate Researcher (Doctor of Sports Nutrition), Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE072415
Record Dates: First submitted 2025-11-28; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Performance Enhancement; Supplemental Nutrition Assistance Program Education; Strength Outcomes; Function Improvement; Intervention Study
Keywords: Multiple sclerosis; Omega-3; nutritional supplements
MeSH Terms: conditions — Multiple Sclerosis | interventions — Docosahexaenoic Acids; Dietary Supplements; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: A randomized parallel study will be conducted in which 100 participants with multiple sclerosis will be divided into four groups: one group will take 2 g of DHA (4 capsules; n = 25), another group will take 2 g of DHA (4 capsules; n = 25) combined with therapeutic exercise, a third group will take placebo (4 capsules; n = 25), and a fourth group will take placebo (4 capsules; n = 25) combined with therapeutic exercise.
  All participants will complete the study. The duration of the intervention will be 3 months.
  DHA = docosahexaenoic acid. Placebo = sunflower oil.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The company that formulated the Omega-3 and placebo carried out the randomization, so no one on the research team or among the sponsors knew which group each study subject belonged to. The results of the randomization were sent to our laboratory after the study was completed to determine which subjects were in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DHA (Experimental): This group will take 2 g of DHA (4 capsules per day) for 3 months
  Interventions: Dietary Supplement: Docosahexaenoic Acid (DHA) Dietary Supplement
- DHA + therapeutic exercise (Experimental): This group will take 2 g of DHA (4 capsules per day) + therapeutic exercise for 3 months
  Interventions: Dietary Supplement: Docosahexaenoic Acid (DHA) Dietary Supplement
- Sunflower oil (Placebo Comparator): This group will take a placebo (4 capsules per day) for 3 months.
  Interventions: Dietary Supplement: Sunflower Oil
- Sunflower oil + therapeutic exercise (Placebo Comparator): This group will take a placebo (4 capsules per day) + therapeutic exercise for 3 months.
  Interventions: Dietary Supplement: Sunflower Oil

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic Acid (DHA) Dietary Supplement — Subjects will take 2 g of DHA per day for 3 months.
  Other Names: Omega-3
  Arms: DHA
Dietary Supplement: Docosahexaenoic Acid (DHA) Dietary Supplement — Subjects will take 2 g of DHA per day + therapeutic exercise (3 times a week) for 3 months.
  Arms: DHA + therapeutic exercise
Dietary Supplement: Sunflower Oil — Subjects will take 2 g of placebo (sunflower oil) per day for 3 months.
  Other Names: Placebo
  Arms: Sunflower oil
Dietary Supplement: Sunflower Oil — Subjects will take 2 g of placebo per day + therapeutic exercise (3 times a week) for 3 months.
  Arms: Sunflower oil + therapeutic exercise

SUMMARY:
This clinical trial will investigate the effects of combining therapeutic exercise with DHA supplementation in 100 patients with multiple sclerosis using a randomized controlled design. Participants, diagnosed according to the McDonald criteria, will undergo functional, cognitive, fatigue, and quality-of-life assessments through tools such as the EDSS, BRB-N, MFIS, EVA-f, and MSQoL-54. Physiological evaluations will include infrared thermography, isokinetic strength testing, perceived exertion (Modified Borg Scale), balance (Timed Up and Go), lower-limb power (Sit-to-Stand app), and handgrip strength. The study hypothesizes that this combined intervention will improve motor function, cognition, fatigue management, and overall quality of life by enhancing neuromuscular activation and metabolic efficiency.

DETAILED DESCRIPTION:
Design

Randomized clinical trial.

Study Period

Two years: from January 2024 to January 2026.

Population Selection Reference Population

The study sample will be recruited from the Multiple Sclerosis Association (AMDEM) in the Region of Murcia and the Neurology Department of Hospital Ribera Salud in Molina de Segura.

Eligible participants will be patients diagnosed with multiple sclerosis (MS) according to the McDonald criteria, aged approximately 18 to 65 years, who have not experienced relapse episodes in the month prior to inclusion, and have an Expanded Disability Status Scale (EDSS) score between 0.0 and 6.0, as well as the ability to voluntarily activate the tibialis anterior muscle.

Sample Size

Given the characteristics of the study, the target sample size is at least 100 participants, divided into four groups (n ≈ 25 per group) according to treatment.

Participants will be randomly assigned to one of four groups, each following a different therapeutic protocol:

Group 1: therapeutic exercise protocol three times per week throughout the study + daily DHA supplementation (4 capsule/day).

Group 2: same exercise protocol + placebo capsule (sunflower oil) identical in appearance, color, and dosage.

Group 3: DHA supplementation only (4 capsule/day).

Group 4: placebo capsule only (sunflower oil), identical to intervention groups.

Statistical Design

A one-way or repeated-measures ANOVA will be used to test for statistically significant differences among three or more dependent samples.

Measurement time points will be defined as follows:

T0: baseline (pre-intervention).

T1: midpoint of the intervention (approximately 1.5 months after initiation).

T2: immediately after completing the 3-month intervention protocol.

T3: 3 months after the end of the intervention.

Data Collection Participant Characteristics

Sensitive data will be collected regarding:

Age, sex, height, weight, medication use, relapse episodes in the months prior to the study, disability status, disease condition, and cognitive function.

Additional psychophysical information will be gathered using validated questionnaires administered before and after the intervention:

Disability will be assessed using the Expanded Disability Status Scale (EDSS).

A score of 0.0 represents normal physical function without disability.

3-4 indicates mild impairment not limiting daily or work activities.

5-6 indicates moderate disability, typically able to walk but requiring assistance for about 100 meters at level 6.

7-9 represents severe impairment, often confined to a wheelchair or bed.

Cognitive function will be assessed using the Brief Repeatable Battery of Neuropsychological Tests (BRB-N), a validated tool for MS. It includes tests of selective recall, the 7/24 spatial recall test, the controlled oral word association test, and the paced auditory serial addition test (PASAT).

Fatigue will be measured using the Modified Fatigue Impact Scale (MFIS), assessing the perceived impact of fatigue on cognitive (10 items), physical (10 items), and psychosocial (20 items) functioning. Responses range from 0 (no problem) to 4 (extreme problem), with a maximum score of 160.

Quality of life will be measured with the Multiple Sclerosis Quality of Life-54 (MSQoL-54), a validated MS-specific scale that evaluates symptom severity, walking ability, absenteeism due to health, hospitalization history, depressive symptoms, and disease duration.

Functional Assessments

Pre, during and post--intervention.

Infrared thermography will capture whole-body thermal images before, during, and after the intervention as a non-invasive, reliable, and cost-effective diagnostic tool. Measurements will be taken:

Pre and post--intervention.

The Modified Borg Scale will be used to adjust exercise load intensity, maintaining perceived exertion between 5-7. If the score falls below 5, resistance will be increased by adding up to 5 kg. This will be recorded in the final session of each week.

The EVA-f scale (adapted fatigue visual analogue scale) will be used to measure subjective fatigue perception (0 = no fatigue; 10 = extreme fatigue) at the end of each training session.

The Sit-to-Stand App Test will be used to assess lower-limb power through video-based analysis of standing-up movements, providing values for time, power, and velocity (pre- and post-protocol).

The Timed Up and Go (TUG) Test will assess balance and fall risk. Participants will stand up from a chair, walk 3 meters, turn around, return, and sit down again. Two repetitions per session will be performed with one-minute rest intervals.

Handgrip strength will be measured (pre- and post-intervention) to assess upper-limb muscle strength.

Isokinetic strength tests will evaluate lower-limb strength (pre- and post-intervention).

Laboratory Tests

Serum analyses will include measurement of interleukin-6,

Blood samples will be collected at four time points:

Pre, during and immediately post-intervention.

ELIGIBILITY:
Inclusion Criteria:

The patient sample comes from the Multiple Sclerosis Association (AMDEM) of the Murcia region and the neurology department of the Ribera Salud Hospital in Molina de Segura. Patients diagnosed with multiple sclerosis according to the McDonald criteria, aged between 18 and 65 (approximately), who have not suffered any flare-ups in the previous month and who have a score of 0.00 to 6 on the Expanded Disability Status Scale (EDSS) and are able to activate the tibialis anterior muscle will be eligible for the study.

Exclusion Criteria:

* Not fulfilling the inclusion criteria.
* Having any problems performing the tests.
* Having any problems taking the supplement or placebo.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
ISOKINETIC | Throughout study completion, an average of 12 weeks
  Measurement of isokinetic strength in the right leg N/m

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale | Throughout study completion, an average of 12 weeks
  Fatigue is assessed using the Modified Fatigue Impact Scale, which considers the perceived impact of fatigue on cognitive functioning (10 items), physical functioning (10 items) and psychosocial functioning (20 items). It is a self-administered instrument in which subjects are asked to rate the extent to which fatigue has caused them problems (0 = no problem to 4 = extreme problem, maximum score = 160).
MSQoL-54 - Walking Status | Throughout study completion, an average of 12 weeks
  Description: Functional walking status assessed using the walking-related item of the MSQoL-54.
  Unit of Measure: Categorical (able to walk without assistance / needs assistance / wheelchair dependent).
MSQoL-54 - Days Unable to Work or Attend School Due to Health | Throughout study completion, an average of 12 weeks
  Description: Number of days participants were unable to work or attend school due to health problems during the previous month, assessed via MSQoL-54.
  Unit of Measure: Days (0, 1-15, 16-30).
MSQoL-54 - Hospital Admission in the Previous Year | Throughout study completion, an average of 12 weeks
  Description: Self-reported hospital admission related to health status in the previous year, assessed via MSQoL-54.
  Unit of Measure: Binary (yes/no).
MSQoL-54 - Depressive Symptoms | Throughout study completion, an average of 12 weeks
  Description: Presence of self-reported depressive symptoms assessed using the corresponding MSQoL-54 item.
  Unit of Measure: Binary (yes/no).
THERMOGRAPHY | Pre, six weeks after the start and after the intervention (12 weeks)
  Thermography study to capture full-body thermal images will be performed using a Flir E75 camera. The temperature (°C) of the lower limbs will be evaluated by analyzing the images.
SIT TO STAND TEST | Throughout study completion, an average of 12 weeks
  The Sit to Stand app test will be performed and muscle power will be assessed using the application. This tool is based on video recording of the movement of getting up from a chair. The unit of measurement is meters/seconds.
TIME UP AND GO test | Throughout study completion, an average of 12 weeks
  The Time Up and Go test will be implemented, which is a method of assessing balance ability consisting of several parts, where the patient starts sitting in a chair, then stands up and walks 3 metres, turns around to return to the chair and then sits down, measuring the time it takes to complete the task. Each measurement will be repeated twice with a one-minute rest in between. To perform this test, the patient needs good posture control, coordination and strength in the lower limbs, and balance, movement control and risk of falls are assessed. The unit of measurement is in seconds.
HAND GRIP | Throughout study completion, an average of 12 weeks
  Hand grip to assess upper limb strength through pre- and post-treatment grip strength. The unit of measurement is the kilogram.
IL-6 | Pre, six weeks after the start and after the intervention (12 weeks)
  Serum interleukin 6 levels will be determined by blood sampling performed by an experienced nurse and analyzed in our reference laboratory.
MSQoL-54 - Multiple Sclerosis Disease Duration | Baseline
  Description: Duration of multiple sclerosis since diagnosis.
  Unit of Measure: Years.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Martínez Noguera, Researcher-PhD, Study Chair — Universidad Católica San Antonio de Murcia
Locations (1):
- Research Center for High Performance Sport. Universidad Católica de Murcia, La Ñora, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research Center for High Performance Sport. Universidad Católica de Murcia. — https://investigacion.ucam.edu/vicerrectorado/ciard